CLINICAL TRIAL: NCT06060652
Title: Prostate Oligometastatic Cancer Management Driven by Disease Biology et/or Immunoactivity (PROMETEO)
Acronym: PROMETEO
Status: Recruiting | Type: Observational
Sponsor: Centro di Riferimento Oncologico - Aviano (Other)
Responsible Party: Sponsor
Other Study IDs: CRO-2023-11
Record Dates: First submitted 2023-09-25; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Oligometastatic Prostate Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective cohort: 34 OMPC patients enrolled in the ADAPT-CTC trial
- Prospective cohort: A minimum sample size of 70 OMPC patients undergoing SBRT must be enrolled in this study to satisfy the study endpoints

SUMMARY:
Currently, despite the advent of next-generation imaging has improved the detection of Oligometastatic prostate cancer (OMPC), prognostic biomarkers able to stratify patients and monitor treatment response are lacking and urgently needed. Mounting evidence suggests that molecular profiling of the disease and host immune activity evaluation can reveal OMPC heterogeneity and address the above unmet clinical need.

This study aims at combining the analysis of several biomarkers to improve the prognostic stratification of OMPC patients

DETAILED DESCRIPTION:
Currently, despite the advent of next-generation imaging has improved the detection of Oligometastatic prostate cancer (OMPC), prognostic biomarkers able to stratify patients and monitor treatment response are lacking and urgently needed. Mounting evidence suggests that molecular profiling of the disease and host immune activity evaluation can reveal OMPC heterogeneity and address the above unmet clinical need.

Liquid biopsy, defined as the sampling and analysis of tumor-derived analytes [i.e.: circulating tumor cells (CTCs), or circulating tumor DNA (ctDNA)] from blood, represents a powerful tool to assess in real-time the evolving landscape of cancer, identify prognostic and predictive biomarkers and detect resistance to therapies in several cancers, including Prostate Cancer (PC).

Additionally, the same blood sample allows the profiling of tumor-associated components, such as circulating immune cells, which may give clues at the systemic level about the dynamic and complex host-tumor interaction. It is non-invasive, easily repeatable, and cost-effective. In this regard, preliminary results derived from clinical studies indicate that the analysis of tumor material circulating in peripheral blood, combined with the study of the host immune response might be pivotal. This study aims at combining the analysis of several biomarkers, associated with both tumor (CTC and cfDNA) and host (TCR), with a micro-invasive approach, such as liquid biopsy, to improve the prognostic stratification of OMPC patients compared to conventional laboratory test (PSA) and imaging exams (Choline- or PSMA-PET imaging).

ELIGIBILITY:
Inclusion criteria

Retrospective cohort

* >18 years old;
* Patients previously included in the ADAPT-CTC trial
* Signing written informed consentInclusion Criteria:

Prospective cohort

* >18 years old
* Histologic confirmation (primary or metastatic tumor) of Acinar Adenocarcinoma of Prostate
* Hormone-sensitive OMPC defined as ≤3 metachronous metastases (bone and/or lymph node) detected within the past 6 months with Choline/PSMA PET-CT following prostate specific antigen (PSA) rising after primary treatment (surgery and/or radiotherapy) with curative intent as defined by European Association of Urology criteria (EAU).
* Controlled primary tumor
* Prior salvage treatment to the primary prostate cancer is allowed.
* PSA ≤ 50 ng/mL
* Testosterone ≥ 0.5 ng/mL
* ADT associated to the primary treatment concluded more than 6 months prior to the enrollment.
* Patients eligible for a course of SBRT on bone and/or lymph node metastatic sites
* Patients must have a life expectancy ≥ 12 months and an ECOG performance status ≤ 2
* Patients must have normal organ and marrow function defined as:

  * Leukocytes ≥2000/µL
  * Absolute Neutrophil Count ≥1000/µL
  * Platelets ≥50000/µL
* Patients amenable to understand and sign written informed consent documents

Exclusion Criteria:

Prospective cohort

* Spinal cord compression or impending spinal cord compression.
* Suspected pulmonary and/or liver metastases
* Patient receiving any other investigational agents
* Patient is participating in a concurrent treatment protocol
* Prior treatments for hormone-sensitive OMPC
* Serum creatinine > 3 times the upper limit of normal.
* Total bilirubin > 3 times the upper limit of normal.
* Liver Transaminases > 5-times the upper limit of normal.
* Unable to lie flat during or tolerate PET/CT or SBRT.
* Previous history of cancer other than non-melanoma skin cancer in the last 5 years
* Traumatic bone events in the 4 weeks before PET

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: OMPC patients undergoing SBRT
Sampling Method: Non-Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2023-05-11 (Actual); Primary Completion 2026-05-11 (Estimated); Study Completion 2026-05-11 (Estimated)

PRIMARY OUTCOMES:
Validation of the prognostic significance of CTCs in a prospective cohort of OMPC patients undergoing SBRT | up to 3 years
  To verify if a cut-off value of ≥5 CTC/7.5 mL of blood is prognostic of worst outcome in terms of distant progression-free survival (DPFS). Prognostic value will be measured as hazard ratio and relative 95% confidence intervals. DPFS will be defined as the time between the first day of SBRT and the detection at restaging imaging of clinical disease outside the treatment field

SECONDARY OUTCOMES:
Biochemical-PSF and CTC | up to 3 years
  Evaluate the relation between CTC number and its variation and biochemical PFS defined as the time between the first day of SBRT to the PSA increase ≥ 25% and ≥ 2 ng/mL if PSA was ≥ 2 ng/mL from baseline, or a PSA increase ≥ 25% if PSA was < 2 ng/mL.
Biochemical-PSF and TCR | up to 3 years
  Evaluate the relation between TCR values and biochemical PFS defined as the time between the first day of SBRT to the PSA increase ≥ 25% and ≥ 2 ng/mL if PSA was ≥ 2 ng/mL from baseline, or a PSA increase ≥ 25% if PSA was < 2 ng/mL.
Identify signatures in cfDNA of prognostic significance in terms of Biochemical-PSF | up to 3 years
  Association between the presence of a combination of specific tumour mutations detected in cfDNA and Biochemical-PSF defined as the time between the first day of SBRT to the PSA increase ≥ 25% and ≥ 2 ng/mL if PSA was ≥ 2 ng/mL from baseline, or a PSA increase ≥ 25% if PSA was < 2 ng/mL.
Distant-PSF and CTC | up to 3 years
  Evaluate the relation between CTC number and its variation and distant PFS defined as the time between the first day of SBRT to the detection at restaging imaging of clinical disease outside the treatment field obtained after biochemical progression
Distant-PSF and TCR | up to 3 years
  Evaluate the relation between TCR values and distant PFS defined as the time between the first day of SBRT to the detection at restaging imaging of clinical disease outside the treatment field obtained after biochemical progression
Identify signatures in cfDNA of prognostic significance in terms of Distant-PSF | up to 3 years
  association between the presence of a combination of specific tumour mutations detected in cfDNA and distant PFS defined as the time between the first day of SBRT to the detection at restaging imaging of clinical disease outside the treatment field obtained after biochemical progression
Local control and CTC | up to 3 years
  Evaluate the relation between CTC number and its variation and local control defined as no evidence of disease in the treatment field at restaging imaging obtained after biochemical progression
Local control and TCR | up to 3 years
  Evaluate the relation between TCR values and local control defined as no evidence of disease in the treatment field at restaging imaging obtained after biochemical progression
Identify signatures in cfDNA of prognostic significance in terms of Local control | up to 3 years
  association between the presence of a combination of specific tumour mutations detected in cfDNA and local control defined as no evidence of disease in the treatment field at restaging imaging obtained after biochemical progression
ADT-free survival and CTC | up to 3 years
  Evaluate the relation between CTC number and its variation and ADT-FS defined as time between the first day of SBRT to the start of palliative ADT
ADT-free survival and TCR | up to 3 years
  Evaluate the relation between TCR values and ADT-FS defined as time between the first day of SBRT to the start of palliative ADT
Identify signatures in cfDNA of prognostic significance in terms of ADT-free survival | up to 3 years
  association between the presence of a combination of specific tumour mutations detected in cfDNA and ADT-FS defined as time between the first day of SBRT to the start of palliative ADT
time to castration resistant Prostate Cancer and CTC | up to 3 years
  Evaluate the relation between CTC number and its variation and TTCR defined as the time between the first day of SBRT to the PSA ≥ 2 ng/mL and Testosterone levels < 0.5 ng/mL
time to castration resistant Prostate Cancer and TCR | up to 3 years
  Evaluate the relation between TCR values and TTCR defined as the time between the first day of SBRT to the PSA ≥ 2 ng/mL and Testosterone levels < 0.5 ng/mL
Identify signatures in cfDNA of prognostic significance in terms of time to castration resistant Prostate Cancer | up to 3 years
  association between the presence of a combination of specific tumour mutations detected in cfDNA and TTCR defined as the time between the first day of SBRT to the PSA ≥ 2 ng/mL and Testosterone levels < 0.5 ng/mL
Overall survival and CTC | up to 3 years
  Evaluate the relation between CTC number and its variation and OS defined as the time between the first day of SBRT to the time of death.
Overall survival and TCR | up to 3 years
  Evaluate the relation between TCR values and OS defined as the time between the first day of SBRT to the time of death.
Identify signatures in cfDNA of prognostic significance in terms of Overall survival | up to 3 years
  association between the presence of a combination of specific tumour mutations detected in cfDNA and OS defined as the time between the first day of SBRT to the time of death.
TCR values | up to 3 years
  Median of TCR diversity, clonality and fold change before and after SBRT
cfDNA | up to 3 years
  Frequency of selected tumour mutations in cfDNA
prognostic value of the combination of different biomarkers | up to 3 years
  difference in distant-PFS probability between subgroups of patients carrying different combination of circulating biomarkers. Distant PFS will be defined as the time between the first day of SBRT to the detection at restaging imaging of clinical disease outside the treatment field obtained after biochemical progression

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Matrone, MD, Principal Investigator — Centro di Riferimento Oncologico (CRO), IRCCS; Giulia Brisotto, PhD, Principal Investigator — Centro di Riferimento Oncologico di Aviano (CRO); Matteo Turetta, MD, Principal Investigator — Centro di Riferimento Oncologico di Aviano (CRO); Fabio Del Ben, MD, Principal Investigator — Centro di Riferimento Oncologico di Aviano (CRO); Luca Triggiani, MD, Principal Investigator — Asst Degli Spedali Civili Di Brescia
Locations (2):
- Italy (2):
  - IRCCS-Centro di Riferimento Oncologico (CRO) di Aviano, Aviano, Pordenone
  - ASST Spedali Civili, Brescia